CLINICAL TRIAL: NCT05700071
Title: Magnetic Resonance Spectroscopy Markers of Glioma Genomics
Brief Title: MRS of Glioma Genomics
Acronym: GLIOMRS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: C21-27; 2021-A03015-36 (Other: IDRCB)
Record Dates: First submitted 2023-01-17; First posted 2023-01-26 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-01

CONDITIONS: Glioma
Keywords: Gliomas; Isocitrate dehydrogenase; 1p19q codeletion; MR Spectroscopy; MRI; Diagnosis; Treatment monitoring
MeSH Terms: conditions — Glioma; Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- MRI examination (Experimental)
  Interventions: Diagnostic Test: MRI

INTERVENTIONS:
Diagnostic Test: MRI — MRI without contrast agent

SUMMARY:
In France, about 5000 new people with a primary malignant brain tumor are diagnosed each year. The most common primary tumors are gliomas, originating from glial cells (astrocytomas and oligodendrogliomas). Low-grade gliomas are mildly aggressive, but they often evolve into a more malignant form.

Mutations in the genes encoding isocitrate dehydrogenase (IDH) are found in about 80% of low-grade gliomas and are associated with a favorable prognosis. Remarkably, IDH-mutated gliomas are characterized by a specific cellular metabolism causing the accumulation of D-2-hydroxyglutarate (2HG) in tumor cells. 2HG can be detected in vivo using 1H magnetic resonance spectroscopy (MRS) and is recognized as a unique, noninvasive biomarker of IDH-mutated gliomas. Noninvasive detection of IDH mutations via 2HG MRS represents a crucial step for decision-making and patient care.

A subset of IDH-mutated tumors also presents a complete deletion of 1p and 19q chromosome arms (1p/19q codeletion). The 1p/19q codeletion is specifically linked to the oligodendroglial histologic subtype and it has been associated with a better patient outcome. However, the biological effects of this genetic alteration are still unclear and in vivo markers are lacking. Recently, we reported the first in vivo detection of the cystathionine molecule in human brain gliomas using MRS and explored the association between cystathionine accumulation and 1p/19q codeletion in gliomas.

In this project, the investigation team will combine cutting edge MRI and MRS techniques for metabolic and microstructural characterization of brain tumors with the aim of providing novel reliable noninvasive biomarkers of tumor genetic subtypes. These methods will enable noninvasive identification of IDH-mutated gliomas and, potentially, 1p/19q codeleted gliomas. In addition, the researchers will investigate the utility of 2HG, cystathionine and MRI microstructural markers to monitor tumor response to anti-cancer treatments and tumor progression.

The outputs of this project, altogether, may open new avenues to a better understanding of the pathophysiological mechanisms of oncogenesis and the design of new treatments for gliomas.

ELIGIBILITY:
Inclusion Criteria:

* Affiliation à un régime de sécurité sociale (bénéficiaire ou ayant droit)
* Recueil du consentement écrit et éclairé
* Une des deux situations suivantes :

Groupe 1 : Probable gliome de grade II/III, dont l'exérèse est programmée

Groupe 2 : gliome de grade II ou III prouvé histologiquement avec statut IDH1/IDH2 connu, n'ayant reçu aucun autre traitement que la chirurgie, et devant débuter un traitement autre que la chirurgie.

* Présence d'un résidu tumoral évaluable (>2 cm de diamètre en FLAIR)
* Index de Karnofsky > 60
* Contraception efficace pendant la durée de la recherche, complété par un test de grossesse négatif pour les femmes en âge de procréer.

Exclusion Criteria:

* Contrindications à l'IRM:

pace maker ou stimulateur neuronal, corps étranger métallique intraoculaire ou intracérébral, implant cochléaire, valve cardiaque ou matériel artériel chirurgical métallique non compatible IRM, matériel métallique susceptible de concentrer les impulsions de radio fréquence, claustrophobie

* femmes enceintes ou allaitantes
* Critères réglementaires :

Femme enceinte, parturiente, allaitante; Absence de signature du consentement ou refus du participant; Mesure de protection juridique (tutelle, curatelle, sauvegarde de justice); Participation à une autre recherche ne permettant pas de respecter la période; d'exclusion entre les 2 recherches; Personne ne bénéficiant pas d'un régime d'assurance maladie

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-03-06 (Actual); Primary Completion 2026-03-03 (Estimated); Study Completion 2028-03-02 (Estimated)

PRIMARY OUTCOMES:
Metabolite concentrations by MRS | 1.5 hour
  Concentrations of 2-hydroxyglutarate and cystahionine measured by MRS will be correlated with IDH mutational status and 1p19q codeletion derived from ex vivo analyses in tumor tissue samples

SECONDARY OUTCOMES:
Diffusion MRI metrics | 1,5 hours
  Diffusion MRI metrics will be correlated with the 1p19q codeletion status derived from ex vivo analyses in tumor tissue samples
Metabolic changes during an anti-tumor treatment | 1 year
  The changes in concentration of 2-hydroxyglutarate, cystathionine and choline will be compared to the changes in tumor volumes and to the clinical response
Diffusion MRI and amide proton transfer signal changes during an anti-tumor treatment. | 1 year
  Diffusion MRI and amide proton transfer signal changes will be compared to the changes in metabolism, tumor volumes and to the clinical response

CONTACTS AND LOCATIONS:
Overall Officials: Francesca Branzoli, PhD, Study Director — Paris Brain Institute, Paris, France; Marc Sanson, MD, PhD, Principal Investigator — Paris Brain Institute, AP-HP, Paris, France
Locations (2):
- France (2):
  - Pitié-Salpetrière Hospital, Paris
  - Hôpital Pitié Salpêtrière, 47 Boulevard de l'Hôpital, 75013 Paris, Paris, Île-de-France Region

IPD SHARING:
Plan to Share IPD: No